CLINICAL TRIAL: NCT07390851
Title: Evaluation of the Effect of Adding Magnesium Sulfate to Lidocaine in the Treatment of Myofascial Pain Dysfunction Syndrome Using Surface Electromyography (sEMG).(Randomized Clinical Trial)
Brief Title: Magnesium Sulfate as an Adjuvant to Lidocaine in MPDS Trigger Point Injections Assessed by VAS and sEMG.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maii Emad Abdelazeem, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-OMFS-MPDS-TP-2025
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Myofascial Pain Dysfunction Syndrome
Keywords: Trigger points injection; Myofascial Pain Dysfunction Syndrome (MPDS); Magnesium Sulfate; Surface Electromyography; Visual Analog Scale
MeSH Terms: conditions — Fibromyalgia | interventions — Lidocaine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups. Group 1 will receive lidocaine trigger point injections, while Group 2 will receive lidocaine combined with magnesium sulfate. Outcomes will be assessed at predefined follow-up visits using VAS and surface EMG.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a randomized single-blinded trial. Participants and outcome assessors are blinded to the injection material. The clinician performing the injections is not blinded due to preparation and administration requirements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine injection (Active Comparator): 2%preservative-free without vasocostrictor injectable solution, 1.8 ml per injection point.
  Interventions: Drug: Lidocaine 2% (preservative-free, without vasoconstrictor)
- Injection of Magnesium sulfate with Lidocaine (Experimental): 10% injectable solution (100 mg/ml), from certified supplier. Approx. 3.8 ml per point (1.8 ml Lidocaine + 2 ml MgSO₄)
  Interventions: Drug: Lidocaine 2% + Magnesium Sulfate 10% (combination)

INTERVENTIONS:
Drug: Lidocaine 2% (preservative-free, without vasoconstrictor) — Using 25-27G sterile disposable needle, intramuscular injection of 2%preservative-free solution of lidocaine without vasocostrictor, 1.8 ml at the most painful trigger points with "Fast-in, fast out" or "peppering" method and inject the solution slowly.
  Arms: Lidocaine injection
Drug: Lidocaine 2% + Magnesium Sulfate 10% (combination) — Using 25-27G sterile disposable needle, intramuscular injection of 2%preservative-free solution of lidocaine without vasocostrictor mixed with 10%magnesium sulphate , Approx. 3.8 ml per point (1.8 ml Lidocaine + 2 ml MgSO₄) at the most painful trigger points with "Fast-in, fast out" or "peppering" method and inject the solution slowly.
  Arms: Injection of Magnesium sulfate with Lidocaine

SUMMARY:
Two groups of patients diagnosed with Myofascial Pain Dysfunction Syndrome (MPDS) will be included in this study. One group will receive trigger point injections of lidocaine alone. The other group will receive trigger point injections of lidocaine combined with magnesium sulfate. The study aims to compare the effectiveness of both treatments in reducing pain and improving muscle function. Patients will be assessed using a pain scale (VAS) and surface electromyography (sEMG) to measure muscle activity.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate whether adding magnesium sulfate to lidocaine in trigger point injections provides better pain relief and muscle relaxation in patients with Myofascial Pain Dysfunction Syndrome (MPDS) compared to lidocaine alone.

Participants diagnosed with MPDS will be randomly assigned into one of two groups:

Group 1 (Control Group): Trigger point injection of lidocaine 2% Group 2 (Intervention Group): Trigger point injection of lidocaine 2% combined with magnesium sulfate 10% Each participant will receive injections in the identified myofascial trigger points. Pain during injection and after injection will be assessed using the Visual Analog Scale (VAS). Muscle activity will be measured using surface electromyography (sEMG) at specific time points during rest and muscle contraction.

The study will compare the changes in pain scores and EMG readings between the two groups to determine whether magnesium sulfate enhances the analgesic and muscle-relaxing effects of lidocaine. The results of this study may help improve treatment strategies for MPDS and provide evidence for using magnesium sulfate as an adjuvant to lidocaine in trigger point injections.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Clinical diagnosis of Myofascial Pain Dysfunction Syndrome (MPDS).
3. Presence of active myofascial trigger points in accessible muscles (e.g., masseter, temporalis, upper trapezius).
4. Pain duration ≥ 3 months.
5. Pain intensity ≥ 4 on the Visual Analog Scale (VAS).
6. Noprior trigger point injection in the affected area within the past 3 months.
7. Ability and willingness to provide informed consent.
8. Compliance with study visits and procedures

Exclusion Criteria:

1. Known allergy or hypersensitivity to Lidocaine, Magnesium Sulfate, or related agents.
2. Current use of anticoagulants or history of bleeding disorders.
3. Systemic or local infection at or near the injection site.
4. History of fibromyalgia, central pain syndromes, or cancer-related pain.
5. Major psychiatric illnesses (e.g., schizophrenia, severe depression).
6. Recent surgery or trauma to the head, neck, or upper back (<6 months).
7. Use of analgesics (NSAIDs, opioids) within 5 days before intervention.
8. Severe systemic diseases:- Uncontrolled diabetes mellitus- Liver or kidney failure- Severe cardiovascular conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Pain reduction. | Baseline, 1week, 2 weeks post-injection.
  Pain intensity will be assessed using the Visual Analogue Scale (VAS) ranging from 0 to 10 cm, where 0 indicates no pain and 10 indicates worst imaginable pain.
Muscle activity improvement. | Baseline, 1 week, 2 weeks post-injection
  Muscle activity will be assessed using surface electromyography (sEMG) by measuring Maximum Voluntary Contraction (MVC) in microvolts (µV). Higher values indicate improved muscle activity.

SECONDARY OUTCOMES:
Pain experienced during injection | Immediately after injection
  Pain during injection will be assessed immediately after injection using the Visual Analogue Scale (VAS) ranging from 0 to 10 cm, where 0 indicates no pain and 10 indicates worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Maii E Abdelazeem, Bsc, Principal Investigator — Faculty of Oral & Dental Medicine, Cairo University
Locations (1):
- Faculty of oral and dental medicine, cairo university, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This is an academic thesis-based study, and the data contain sensitive personal and clinical information. Data access is restricted by institutional policies and ethical approval requirements. De-identified aggregate results will be reported in publications.

REFERENCES:
- [Background] Leitch J, Webb A, Pudwell J, Chamberlain S, Henry R, Nitsch R. Magnesium-Based Trigger Point Infiltrations Versus Local Anaesthetic Infiltrations in Chronic Pelvic Myofascial Pain: A Randomized, Double-Blind, Controlled Study. J Obstet Gynaecol Can. 2022 Aug;44(8):877-885. doi: 10.1016/j.jogc.2022.02.129. Epub 2022 Mar 24. PMID 35339694
- [Background] Refahee SM, Mahrous AI, Shabaan AA. Clinical efficacy of magnesium sulfate injection in the treatment of masseter muscle trigger points: a randomized clinical study. BMC Oral Health. 2022 Sep 19;22(1):408. doi: 10.1186/s12903-022-02452-3. PMID 36123724